CLINICAL TRIAL: NCT03731598
Title: The Role of Ceramides in Skeletal Muscle
Brief Title: Ceramides in Muscle During Insulin Resistance
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty recruiting. Objectives from this protocol added to another protocol collecting the same information.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Associate Professor, University of Utah
Other Study IDs: DK115824
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Bed Rest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect blood and muscle biopsy specimens before (Day 1 bed rest) and after bed rest (Day 5 bed rest)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bed rest — Volunteers will be physically inactive on bed rest at the clinical research center

SUMMARY:
Overnutrition and physical inactivity promote the accumulation of sphingolipids such as ceramides which block insulin signaling and anabolic metabolism. Implementation of pharmacological or genetic interventions to reduce sphingolipid levels in rodents prevents or reverses an impressive array of metabolic pathologies (e.g. insulin resistance, diabetes, steatohepatitis, hypertension, cardiomyopathy, and atherosclerosis). To elucidate the tissue-specific mechanisms through which ceramides contribute to these diseases, mice have been produced to allow for the conditional, cell-type restricted ablation of enzymes required for ceramide biosynthesis or degradation (i.e. serine palmitoyltransferase and dihydroceramide desaturases-1) or degradation (i.e. acid ceramidase). Aims of the project include the following: To use these novel mouse models to evaluate the effect of muscle-specific ceramide depletion or induction on insulin sensitivity, muscle growth, and genomic/proteomic signatures under conditions of overnutrition and inactivity. To apply a ceramide flux assay in isolated human myotubes to identify the regulatory mechanisms that influence rates of ceramide biosynthesis; and, To determine the efficacy of a new class of inhibitors of dihydroceramide desaturases-1, our preferred target in the ceramide synthesis pathway, as therapeutics that improve muscle insulin sensitivity and prevent muscle loss in rodents. Findings obtained from these studies could uncover new nutrient-sensing machinery that modulates insulin sensitivity and muscle growth. Moreover, the translational component could lead to new pharmacological approaches for improving muscle health.

DETAILED DESCRIPTION:
Healthy, insulin sensitive, physically active male and female adults will be studied (N=15; 65-80 years as determined by sample size calculation below) recruited from the Salt Lake City area. Inclusion and exclusion criteria can be found in Protection of Human Subjects. Outpatient blood screening, including an oral glucose tolerance (OGTT) test, and bed rest experiments will take place in the University Center for Clinical and Translational Sciences (CCTS), a clinical service supported by an NIH Clinical and Translational Science Award. The CCTS medical supervising physician oversees procedures. Participants will arrive at the CCTS fasted on Day 1 and a euglycemic-hyperinsulinemic clamp study will be performed as done previously with this unit. Vastus lateralis muscle biopsies will be obtained before and three hours after the clamp. Periodic blood samples will be obtained as part of the clamp procedure for measurement of insulin and glucose. Muscle samples will be either cultured or flash-frozen in liquid nitrogen and stored for later analysis. After completion of the first insulin clamp experiment (Day 1), subjects will adhere to 5-days of strict bed rest as this is a clinically-relevant time frame for older adults hospitalized for acute medical illness, as well as being sufficient to induced insulin resistance. Established safety and comfort guidelines will be followed as done previously. On Day 5, after an overnight fast, a second insulin clamp study will be conducted and muscle biopsies will be again obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 60 yrs and older
2. Ability to sign informed consent
3. Free-living, prior to admission

Exclusion Criteria:

1. Cardiac abnormalities considered exclusionary by the study physician
2. Uncontrolled endocrine or metabolic disease (e.g., hypo/hyperthyroidism, diabetes)
3. Globular filtration rate <65 mL/min/1.73m2 or evidence of kidney disease or failure
4. Vascular disease or risk factors of peripheral atherosclerosis. (e.g., uncontrolled hypertension, obesity, diabetes, hypercholesterolemia > 250 mg/dl, claudication or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal and pedal arteries)
5. Risk of deep vein thrombosis including family history of thrombophilia, deep vein thrombosis, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocysteinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombin III
6. Use of anticoagulant therapy (e.g., Coumadin, heparin)
7. Elevated systolic pressure >150 or a diastolic blood pressure > 100
8. Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
9. Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
10. Inability to abstain from smoking for duration of study
11. A history of > 20 pack per year smoking
12. HIV or hepatitis B or C
13. Recent anabolic or corticosteroids use (within 3 months)
14. Subjects with hemoglobin or hematocrit lower than accepted lab values
15. Agitation/aggression disorder (by psychiatric history and exam)
16. History of stroke with motor disability
17. A recent history (<12 months) of gastrointestinal bleed
18. Liver disease
19. Respiratory disease (acute upper respiratory infection, history of chronic lung disease with resting oxygen saturation <97% on room air)
20. Any other condition or event considered exclusionary by the PI and faculty physician

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older community dwelling participants in salt lake city and surrounding cities
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | Change in glucose infusion rate at Day 5 of bed rest (from Pre bed rest)
  Steady state glucose infusion rate in response to constant insulin will be determined by a 3-hour hyperinsulinemic-euglycemic clamp procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Summers, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - The University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
We will provide access to all data collected as a part of this research. Investigators may request access to the shared data generated by this study. All external investigators must submit a written request identifying the research question they are examining and specifying the data they are interested in receiving. The request must include a data security plan and explanation of how the data will be stored and who will have access to the data. All requests will be reviewed by Drs. Summers and Drummond to be sure appropriate NIH requirements are followed.